CLINICAL TRIAL: NCT06643247
Title: The Regulatory Mechanisms of Electroacupuncture Intervention on Immune Cells in Herpes Zoster
Brief Title: Electroacupuncture Regulation of Immune Cells in Herpes Zoster
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Yan Shi, Director, First People's Hospital of Hangzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZN-2024349-01
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Herpes Zoster; Electroacupuncture; Immune
MeSH Terms: conditions — Herpes Zoster | interventions — Pharmaceutical Preparations; Dosage Forms; Electroacupuncture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug group (Active Comparator): Control group
  Interventions: Drug: Drug
- Drugs combined with electroacupuncture group (Experimental): Observation group
  Interventions: Drug: Drug; Procedure: Electroacupuncture

INTERVENTIONS:
Drug: Drug — 1) Valacyclovir Hydrochloride tablets, 0.3 g per dose, twice daily; 2) Mecobalamin tablets, 0.5 mg, three times daily. Taken continuously for 7 days.The affected skin is kept clean and protected to maintain lesion integrity.
  Other Names: Medication
Procedure: Electroacupuncture — Electroacupuncture Treatment: Needling acupoints include the Jiaji points corresponding to the spinal nerve segment of the affected area, Ashi acupoints along the affected zone, and bilateral Hegu and Waiguan points. Electroacupuncture will be performed once daily for 30 minutes per session, with a total of 7 consecutive sessions. The Jiaji and Ashi acupoints will be connected to an electroacupuncture device, set to disperse-dense wave stimulation at a frequency of 2/100 Hz, with current intensity adjusted to the patient's tolerance level.
  Other Names: EA
  Arms: Drugs combined with electroacupuncture group

SUMMARY:
Herpes Zoster (HZ), caused by the Varicella-Zoster Virus (VZV), is a common infection characterized by localized pain and blistering, with higher incidence in females. HZ affects patients' physical health, mental well-being, and quality of life. The immune system is critical in HZ pathogenesis. Studies show acupuncture relieves pain, modulates immunity, and may lower postherpetic neuralgia (PHN) risk. However, evidence is limited on whether electroacupuncture (EA) alleviates HZ by modulating immune cells. Using mass cytometry (CyTOF), this study will analyze peripheral immune cell changes pre- and post-EA to explore its regulatory effects on HZ immunity. This study will recruit HZ patients and healthy controls (HC), dividing patients into medication-only and medication+EA groups to assess EA's potential immunomodulatory effects in HZ treatment.

DETAILED DESCRIPTION:
The study will enroll 8 HZ patients who meet the inclusion criteria and 3 age- and gender-matched healthy controls (HC). HZ patients will be randomly assigned in a 1:1 ratio to a medication-only group or a medication plus electroacupuncture group. All participants will receive Valacyclovir Hydrochloride tablets and Mecobalamin tablets. HZ-related immune cells in peripheral blood will be analyzed using CyTOF before treatment (day 0), during treatment (day 4), and after treatment (day 7). Pain intensity and characteristics will be assessed using the Visual Analogue Scale (VAS) and the Douleur Neuropathique 4 (DN4) questionnaire. Lesion healing (time to vesicle cessation, crusting, and scab detachment) and adverse events will also be recorded to evaluate lesion regression in HZ patients.

ELIGIBILITY:
Inclusion Criteria for HZ:

* Meets HZ diagnostic criteria;
* Female, aged between 50 and 70 years;
* Disease duration ≤7 days, with no prior antiviral, analgesic, or other treatments;
* Herpetic lesions limited to the trunk, within 1 to 3 dermatomes;
* Willing to participate in the trial and has signed the informed consent form.

Inclusion Criteria for HC:

* No history of HZ or major cardiovascular, respiratory, digestive, urinary, hematologic, endocrine, or neurological diseases;
* Age-matched female HC volunteers for the HZ group;
* Clear consciousness and ability to communicate normally;
* Fully understands the study protocol, demonstrates good compliance, and is willing to cooperate with the study;
* Has signed a written informed consent form.

Exclusion Criteria:

* Special types of herpes zoster, including ophthalmic, otic, visceral, meningeal herpes zoster, and zoster sine herpete;
* Women who are planning to conceive, pregnant, or breastfeeding;
* Patients with severe primary diseases of the circulatory, respiratory, or endocrine systems, or systemic failure;
* Patients with bleeding tendencies;
* Use of corticosteroids or immunosuppressants within the past month.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood immune cell levels | Before (Day 0), during (Day 4) and after (Day 7) treatment.
  1. Custom Detection Panel: A 42-color detection panel is specifically designed according to the study objectives and target cell subpopulations. 2. Sample Collection and Processing: Peripheral blood (5 ml) is collected from patients into EDTA purple-top anticoagulant tubes, stored/transported at 4°C, and processed within 48 hours using Ficoll to isolate the PBMC layer, yielding a single-cell suspension of PBMCs. PBMCs can be cryopreserved for batch analysis or processed fresh for immediate analysis. 3. Staining and Analysis: Samples are stained and analyzed over two days. Surface antibodies are stained on the first day, followed by membrane permeabilization and intracellular antibody staining on the second day, before proceeding with CyTOF analysis.

SECONDARY OUTCOMES:
Visual Analogue Scale | Before treatment (Day 0) and after each treatment (Day 1- Day 7).
  The Visual Analogue Scale (VAS) is used to assess pain and is widely applied in clinical practice in China. The basic method involves a 10 cm sliding ruler with one side marked with 10 increments. One end is labeled "0," indicating no pain, and the other end is labeled "10," representing the most intense, unbearable pain.
Douleur Neuropathique 4 questions | Before treatment (Day 0) and after each treatment (Day 1- Day 7).
  The DN4 questionnaire consists of 10 items, with 7 items describing symptoms and 3 items related to clinical examination. Symptom descriptions include burning pain, cold pain, electric shock pain, tingling, pins and needles, numbness, and itching. Clinical examination includes decreased touch sensation, decreased pinprick sensation, and whether brushing in the painful area triggers or increases pain. Each item has "Yes" and "No" options, with "Yes" scored as 1 and "No" scored as 0, for a total score of 10. A score of ≥4 indicates a diagnosis of neuropathic pain.
Lesion Regression Time | Before treatment (Day 0) and after each treatment (Day 1- Day 7).
  The time for blister cessation, crusting, and scab shedding is recorded.
Occurrence of adverse reactions | During the intervention.
  Record the occurrence of adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No